CLINICAL TRIAL: NCT05469386
Title: Single and Combined Effects of Positive Behavior Support, Medication and Academic Accommodation for Children With ADHD
Brief Title: Single and Combined Effects of Behavioral, Academic, and Medication Treatments for ADHD in the Classroom
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 800013424
Record Dates: First submitted 2022-07-14; First posted 2022-07-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo capsule administered in the morning
  Interventions: Behavioral: Behavioral classroom; Behavioral: General Classroom; Behavioral: Academic Accommodations
- Methylphenidate ER (.3 mg/kg dose) (Experimental): Methylphenidate ER (.3 mg/kg dose)administered in the morning
  Interventions: Behavioral: Behavioral classroom; Behavioral: General Classroom; Behavioral: Academic Accommodations
- General Classroom (Active Comparator): General classroom procedures
  Interventions: Drug: Methylphenidate Hydrochloride ER; Drug: Placebo; Behavioral: Academic Accommodations
- Positive Behavior Support Classroom (Experimental): Positive Behavior Support Classroom procedures
  Interventions: Drug: Methylphenidate Hydrochloride ER; Drug: Placebo; Behavioral: Academic Accommodations
- Academic accommodations (Experimental): Academic accommodations are used during seat work and quiz
  Interventions: Drug: Methylphenidate Hydrochloride ER; Behavioral: Behavioral classroom; Drug: Placebo; Behavioral: General Classroom

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride ER — Methylphenidate Hydrochloride ER (.3 mg/kg dose q.d.)
  Arms: Academic accommodations; General Classroom; Positive Behavior Support Classroom
Behavioral: Behavioral classroom — Enhanced positive behavior supports implemented in classroom
  Arms: Academic accommodations; Methylphenidate ER (.3 mg/kg dose); Placebo
Drug: Placebo — Placebo capsule
  Arms: Academic accommodations; General Classroom; Positive Behavior Support Classroom
Behavioral: General Classroom — General education classroom procedures
  Arms: Academic accommodations; Methylphenidate ER (.3 mg/kg dose); Placebo
Behavioral: Academic Accommodations — Accommodations are introduced to support the child's independent seat work completion and quiz scores
  Arms: General Classroom; Methylphenidate ER (.3 mg/kg dose); Placebo; Positive Behavior Support Classroom

SUMMARY:
This study is the first to systematically evaluate the efficacy of single and combined academic accommodation, behavioral treatment, and medication treatment in a large sample of children with ADHD. Using a scientifically rigorous, cross-over design the impact of these approaches on ecologically valid measures of outcome (on-task behavior, quiz scores, academic productivity) will be assessed to inform effective school intervention.

ELIGIBILITY:
Inclusion Criteria:

* ADHD Diagnosis
* IQ >= 70

Exclusion Criteria:

* Prior adverse reaction to methylphenidate
* Autism Spectrum disorder level 2/3
* Child is home schooled

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral frequency count of rule violations | Through study completion, a maximum of eight weeks
  Behavioral frequency count of rule violations. Lower scores are better.
Seatwork completion | Through study completion, a maximum of eight weeks
  Percentage of assigned seat work items completed correctly. Range of scores is from 0-100%. Higher scores are better.
Quiz Scores | Through study completion, a maximum of eight weeks
  Percentage correct out of 10 quiz questions. Range of scores is from 0-100%. Higher scores are better.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - FIU Center for Childern and Families, Miami, Florida
  - Center for Children and Families, Amherst, New York